CLINICAL TRIAL: NCT00867412
Title: Randomized Study of PET/CT in Pre-Operative Staging of Lung Cancer
Brief Title: Randomized Study of Positron Emission Tomography - Computed Tomography (PET/CT) in Pre-Operative Staging of Lung Cancer
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other); Danish Centre for Health Technology Assessment (Other)
Responsible Party: Ulrik Lassen, MD., PH.D, Rigshospitalet
Other Study IDs: PERALUST
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2009-03-23 (Estimated); Status verified 2009-03

CONDITIONS: Non-Small Cell Lung Cancer; Thoracotomy
Keywords: NSCLC; PET/CT; Surgery; FDG; staging
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conventional staging: Staging with CT, mediastinoscopy and bronchoscopy
- Conventional staging and PET/CT: Staging with CT, mediastinoscopy and bronchoscopy, and PET/CT performed prior to mediastinoscopy

SUMMARY:
Patients with possible operable non-small cell lung cancer are randomised to conventional staging, or conventional staging and PET/CT. According to, patients with operable tumor will be referred to surgery, and the number of thoracotomies and futile thoracotomies wil be compared with the two groups in order to asses the possible benefit of PET/CT.

DETAILED DESCRIPTION:
Patients with possible operable NSCLC after staging with CT are randomised to PET-CT with FDG or not, prior to mediastinoscopy. All patients are referred to mediastinoscopy unless a positive FDG uptake results in a positive biopsy suggesting stage IV disease.

Biopsies are performed according to the following criteria:

1. Lymph nodes are numbered according the Mountain classification, and abnormal lesions must be confirmed histologically, by mediastinoscopy or thoracotomy.
2. PET-positive lesions in the liver must be biopsied unless ultrasound or MRI unequivocally indicate the lesions are benign cysts or haemangioma.
3. PET-negative adrenal lesions are accepted without biopsy if CT scan indicate the lesion is a benign adenoma.
4. PET-positive bone lesions must be evaluated by plain x-ray, CT, MRI, or bone scintigraphy. In case of equivocal findings a biopsy must be performed.
5. PET-positive brain lesions must be confirmed by CT or MRI.

Number of patients:

Patients with clinically operable NSCLC after CT-staging are included. All patients must have mediastinoscopy performed.

All patients referred to mediastinoscopy can be randomised after informed consent. A total of 430 consecutive, non-selected patients are planned. It is anticipated that approximately 60% of the referred patients with clinical stage I-IIIa NSCLC will undergo thoracotomy, and a risk of type I and II error of 5% and 10%, respectively, is accepted. Thus a total of 215 patients are randomised in each arm in order to observe an absolute difference of 15% in the number of thoracotomies. This number seems to be sufficient to evaluate differences in the secondary endpoints.

After inclusion of a total of 220 patients, corresponding to 110 PET-scans, an interim analyses are performed. In case of a highly significant difference in the number of thoracotomies (p < 0,001) the study will be closed.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically operable NSCLC after CT
2. Fit for thoracotomy and lobectomy or pneumectomy after lung function tests
3. CT-scan of thorax, including liver and adrenals with no signs of distant metastases.
4. No medical condition contraindication surgery.
5. Age 18-80
6. No claustrophobia.
7. Negative pregnancy test.
8. No diabetes mellitus.
9. Signed informed consent.

Exclusion Criteria:

1. Radiologically M1 disease.
2. Pregnancy
3. Known claustrophobia.
4. Estimated FEV1 < 30% of expected after surgery.
5. Diabetes mellitus.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2002-01; Primary Completion 2007-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Number of futile thoracotomies | Within 1 year

SECONDARY OUTCOMES:
Number of thoracotomies and survival | Within 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- PET & Cyclotron Unit, Rigshospitalet,, Copenhagen, Denmark

REFERENCES:
- [Derived] Fischer BM, Mortensen J, Hansen H, Vilmann P, Larsen SS, Loft A, Bertelsen AK, Ravn J, Clementsen P, Hoegholm A, Larsen KR, Dirksen A, Skov BG, Krasnik M, Hojgaard L, Lassen U. Multimodality approach to mediastinal staging in non-small cell lung cancer. Faults and benefits of PET-CT: a randomised trial. Thorax. 2011 Apr;66(4):294-300. doi: 10.1136/thx.2010.154476. Epub 2010 Dec 17. PMID 21169287
- [Derived] Fischer B, Lassen U, Mortensen J, Larsen S, Loft A, Bertelsen A, Ravn J, Clementsen P, Hogholm A, Larsen K, Rasmussen T, Keiding S, Dirksen A, Gerke O, Skov B, Steffensen I, Hansen H, Vilmann P, Jacobsen G, Backer V, Maltbaek N, Pedersen J, Madsen H, Nielsen H, Hojgaard L. Preoperative staging of lung cancer with combined PET-CT. N Engl J Med. 2009 Jul 2;361(1):32-9. doi: 10.1056/NEJMoa0900043. PMID 19571281